CLINICAL TRIAL: NCT02605928
Title: INJ-INAR-01 Use of BIP-Needles in Rheumatologic Injections
Brief Title: Use of BIP-Needles in Rheumatologic Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Injeq Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INJ-INAR-01
Record Dates: First submitted 2015-11-12; First posted 2015-11-17 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2016-12

CONDITIONS: Intra-articular Injections
Keywords: Arthritis; Bioimpedance; Glucocorticoid; Intra-articular injection; Needle Guidance
MeSH Terms: conditions — Arthritis | interventions — Needles

ARMS (1):
- BIP Needle (Experimental): Injeq Bioimpedance Probe (BIP) Needle is an injection needle that has bioimpedance measurement capability. It measures bioimpedance and detects synovial fluid during inta-articular injection.
  Interventions: Device: Injeq Bioimpedance Probe (BIP) Needle

INTERVENTIONS:
Device: Injeq Bioimpedance Probe (BIP) Needle — Injeq Bioimpedance Probe (BIP) Needle is an injection needle that has bioimpedance measurement capability. It consists of traditional needle cannulae and removable bioimpedance probe which enables the measurement of bioimpedance. The needle is connected to measurement device and tissue identifying algorithm. Bioimpedance is measured during the operation and the algorithm detects when the needle tip is in contact with synovial fluid.

SUMMARY:
The study focuses on needle guidance in rheumatologic operations - glucocorticoid injections inside joint capsules specifically. The main purpose of the study is to assess and validate the clinical feasibility and performance of Bioimpedance Probe (BIP) Needles and assess the benefits, drawbacks and risks related to use of the BIP Needles.

DETAILED DESCRIPTION:
Clinical device investigation

ELIGIBILITY:
Inclusion Criteria:

* Adult patients having an inflammatory rheumatic disease requiring an intra-articular glucocorticoid injection.

Exclusion Criteria:

* Exclusion criteria are the same as generally for intra-articular glucocorticoid injections (e.g. bacterial infection or recent surgical operation relating the joint).
* In addition for not giving (or not capable to give) the consent personally for any reason is an absolute exclusion criterion.
* In addition pregnant women are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riitta Luosujärvi, PhD MD, Principal Investigator — Helsinki University Hospital, Clinic of Rheumathology
Locations (1):
- Helsinki University Hospital, Clinic of Rheumathology, Helsinki, HUS, Finland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First punctures were utilized for tissue detection model validation and tuning. In pivotal phase, the model kept unchanged. Performance of the device was evaluated from pivotal phase results.
Units Other Than Participants: Injected joints
Period: Overall Study
Arm/Group | BIP Needle
Started | 79; 132 Injected joints
Pivotal Phase, Statistical Phase (First punctures utilized for model tuning. Performance of the device was evaluated after tuning.) | 51; 80 Injected joints
Completed (Included to statistical analysis) | 46; 72 Injected joints
Not Completed | 33; 60 Injected joints
Not completed — Model tuning phase | 28
Not completed — Lack of Efficacy | 5

BASELINE CHARACTERISTICS:
Population: Same patient achieved intra-articular injection to one one or to multiple joints
Arm/Group | BIP Needle
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: years] | 51 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: True Positive Detection of Synovial Fluid Marked in Case Report Form
Description: Measurement device indicates with a sound and visual feedback when needle is in contact with synovial fluid. Physician verifies the location with ultrasound imaging, aspiration of synovial fluid and/or lack of resistance in glucocorticoid injection. Even if the device does not detect the synovial fluid, physician performs the injection when needed. Physician marks to the case report form whether the device provided detections during the puncture and were the detections true or false detections.
Time Frame: During intra-articular injection
Measure: Number (95% Confidence Interval); unit: percentage of injected joints
Units Other Than Participants: Injected joints
Arm/Group | BIP Needle
Number analyzed (Participants) | 46
Number analyzed (Injected joints) | 72
percentage of injected joints | 86 [75 to 93]

ADVERSE EVENTS:
Arm/Group | BIP Needle
Serious Adverse Events (participants affected / at risk) | 0/79
Other Adverse Events (participants affected / at risk) | 2/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIP Needle (N=79)
Painful intra-articular injection (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No